CLINICAL TRIAL: NCT02671123
Title: Evaluation of Effect of Co-registration Between Optical Coherence Tomography (OCT) and Coronary Angiography Onto OCT Guided Percutaneous Coronary Intervention (PCI)
Brief Title: Does Co-registration of OCT and Angiography Reduce Geographic Miss of Stent Implantation?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Francis Hospital, New York (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Principal Investigator, Richard A. Shlofmitz, MD, Chairman of Cardiology- Principal Investigator, St. Francis Hospital, New York
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-02
Record Dates: First submitted 2016-01-26; First posted 2016-02-02 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coronary PCI with OCT with Co-Registration (Active Comparator): Coronary stenting will be performed with OCT guidance as per local practice. Pre and post stenting procedure will be performed with OCT guidance with the use of the Co-Registration software tool after stent implanted.
  Interventions: Procedure: Coronary PCI with OCT with Co Registration
- Coronary PCI with OCT without Co-Registration (Placebo Comparator): Coronary stenting will be performed with OCT guidance as per local practice. Pre and post stenting procedure will be performed with OCT guidance without the use of the Co-Registration software tool after stent implanted.
  I
  Interventions: Procedure: Coronary PCI with OCT without Co Registration

INTERVENTIONS:
Procedure: Coronary PCI with OCT with Co Registration — Co-Registration is an online tool used to take measurements during a stent procedure ( PCI-percutaneous coronary intervention) as part of the OCT ( Optical Coherence Tomography intravascular system. Co Registration software may provide additional imaging details during stent implantation when using OCT.
  Arms: Coronary PCI with OCT with Co-Registration
Procedure: Coronary PCI with OCT without Co Registration — Coronary PCI will be performed using OCT ( Optical Coherence Tomography intravascular system) guidance without the Co Registration software tool enabled.
  Arms: Coronary PCI with OCT without Co-Registration

SUMMARY:
The purpose of this study is to determine whether co-registration of OCT and angiography reduce geographic miss defined as stent edge dissection or significant residual stenosis at stent edge after stent implantation during percutaneous coronary intervention.

DETAILED DESCRIPTION:
Background: When a stent fails to fully cover the lesion, it is termed "geographic miss" (GM). Optical coherence tomography (OCT) is an intracoronary imaging modality that has higher resolution than conventional intracoronary ultrasound. Although OCT allows identification of the location of the culprit lesion and side branch using automated measures, it is sometimes difficult to identify the exact segment corresponding to angiography. Recently, co-registration of OCT and angiography has become available; however, whether this reduces the incidence of GM during stenting is unknown.

Hypothesis: OCT reduces GM during percutaneous coronary intervention.

Objectives:

1. Determine the incidence of GM defined as residual disease* and significant edge dissection† at proximal and distal reference
2. Determine the incidence of stent dislocation (distance between planned and actual stented place)
3. Determine procedural findings (additional stent, total fluoro time, total contrast volume)

   * Minimum lumen area <4.0 mm2 in the presence of significant residual plaque within 5 mm distal and proximal to the stent edge.

     * A flap of vessel wall of >60° is seen in ≥2 consecutive cross-section image within 5 mm distal and proximal from stent edge Study Design and Methods: Single-center, prospective, randomized study. Consented subjects who are to undergo percutaneous coronary intervention are divided into 2 groups randomly (OCT with co-registration vs OCT without co-registration). After stent deployment guided by OCT, dissection, residual disease at the stent edge, and distance between planned and actual stent location are assessed using OCT or angiography. Additional stent deployment, procedure time, total fluoroscopy time, and total contrast volume are also evaluated.

Sample size considerations: OCT with co-registration: 100, OCT without co-registration: 100 (α＝0.05, β ＝0.2). In a retrospective evaluation, the incidence of residual disease (lumen area <4.0 mm2 in the presence of significant residual plaque) or significant stent edge dissection was 36% (18/50, 34% [17/50] with residual stenosis, 4% [2/50] with significant edge dissection). Under the assumption that GM occurs in 36% of patients without co-registration and 18% of patients with co-registration, a group of 190 patients yields a power 80% (with a 2-sided α=0.05) to detect a difference in GM between patients with and without co-registration. In order to account for patient drop out and non-evaluable OCT recordings (5%), a total of 200 patients will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

• Patients ≥18 years old who undergo percutaneous coronary intervention per clinical indications.

Exclusion Criteria:

* Left main disease
* Ostial lesion at Right Coronary Artery
* Tortuous artery in which OCT is unable to pass
* Lesion at bypass graft
* In-stent restenosis
* Chronic total occlusion
* Cardiogenic shock (sustained [>10 min] systolic blood pressure <90 mm Hg in absence of inotropic support or the presence of an intra-aortic balloon pump)
* Acute phase heart failure
* Sustained ventricular arrhythmias
* Known ejection fraction <35%
* Known severe valvular heart disease Known severe renal insufficiency (estimated glomerular filtration rate <30 mL/min/1.72 m2)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Geographic miss | Intraoperative
  Geographic miss defined as evidence of residual disease at stent edge or significant edge dissection after stent deployment

SECONDARY OUTCOMES:
Number of participants with Residual disease at stented edge | Intraoperative
  Residual disease at stent edge will defined as minimum lumen area within 5mm from the stent edge evaluated by OCT. This measurement will be analyzed by a core lab independently who will be blinded for randomization.
Number of participants with stent edge dissection | peri procedure
  Stent edge dissection will be defied as a flap of vessel wall and further categorized as intimal dissection, medial dissection, intramural hematoma, or extra-medial dissection. Minimum lumen area, angle of dissection flap, and length of dissection will be measured by OCT by a core lab who is blinded to the randomization.
Distance between the planned and actual stent location | Intraoperative
  Distance between the planned and actual stent location will be defined as the distance between the center of planned stent location and the center of actual stent location which will be recorded on the OCT software and analyzed by a core lab who is blinded to the randomization.
Number of additional stents required | Intraoperative
  This will be measured as number of participants with additional stent required.
Procedure time | Intraoperative
  time of PCI procedure defined as time vascular access obtained until guide catheter removed from access site.
Total fluoroscopy time | intraoperative
  total amount of fluoroscopy time used during procedure
Total contrast volume | intraoperative
  total mount of contrast in ml used during entire PCI procedure

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Shlofmitz, MD, Principal Investigator — Chairman of Cardiology St Francis Hospital
Locations (1):
- St. Francis Hospital, Roslyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Presently not a plan to share data